CLINICAL TRIAL: NCT00002846
Title: TREATMENT OF METASTATIC RENAL CELL CARCINOMA WITH LOW-DOSE INTRAVENOUS RECOMBINANT INTERLEUKIN-2
Brief Title: Interleukin-2 in Treating Patients With Metastatic or Recurrent Kidney Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Blumenthal Cancer Center at Carolinas Medical Center (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000065085; CMC-09-95-15B; NCI-V96-1038
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2003-12

CONDITIONS: Kidney Cancer
Keywords: stage IV renal cell cancer; recurrent renal cell cancer
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — aldesleukin

INTERVENTIONS:
Biological: aldesleukin
Procedure: conventional surgery

SUMMARY:
RATIONALE: Interleukin-2 may stimulate a person's white blood cells to kill kidney cancer cells.

PURPOSE: Phase II trial to study the effectiveness of low-dose interleukin-2 in treating patients with metastatic or recurrent kidney cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Assess the response rate and survival of patients with metastatic renal cell carcinoma treated with low-dose intravenous interleukin-2.
* Assess the toxicity associated with this treatment.

OUTLINE: Patients receive low-dose intravenous interleukin-2 every 8 hours for a maximum of 15 doses in week 1 and again in week 3. Stable and responding patients receive a second course beginning approximately 2 months after initiation of the first course. Responding patients may continue therapy every 2 months provided toxicity is limited.

Patients whose diseased kidney comprises the bulk of the tumor burden at entry undergo nephrectomy.

Patients are followed for survival.

PROJECTED ACCRUAL: A total of 14 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed renal cell carcinoma (RCC) that is metastatic or recurrent

  * No central nervous system or major nerve involvement
  * No more than 25% estimated hepatic replacement by tumor on CT or MRI
* Measurable disease required

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 80%-100%

Life expectancy:

* Greater than 3 months

Hematopoietic:

* Platelet count at least 80,000/mm3

Hepatic:

* Bilirubin normal
* AST and ALT no greater than 3 times normal

Renal:

* Creatinine normal

Cardiovascular:

* Stress cardiac exam normal (exam performed in patients aged 50 and older and in those with potential cardiac disease suggested by history, physical exam, or EKG)

Pulmonary:

* FEV1 and VC greater than 65% of predicted (tests performed in patients with significant smoking history and in those with potential pulmonary disease suggested by history, physical exam, or x-ray)

Other:

* No sites of ongoing bleeding
* No HIV antibody or AIDS
* No hepatitis B antigen
* No systemic infection
* No requirement for steroids
* No psychiatric disease that precludes informed consent or safe administration of immunotherapy
* No second malignancy except:

  * Basal cell carcinoma
  * In situ cervical cancer
  * Other cancer provided all evaluable lesions are documented RCC
* No pregnant or nursing women
* Effective contraception required of fertile women

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior interleukin-2 therapy

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* At least 28 days since therapy for RCC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 1995-09

CONTACTS AND LOCATIONS:
Overall Officials: Richard L. White, MD, Study Chair — Blumenthal Cancer Center at Carolinas Medical Center
Locations (1):
- Carolinas Medical Center, Charlotte, North Carolina, United States